CLINICAL TRIAL: NCT00512122
Title: Impact of Early Parenteral Nutrition Completing Enteral Nutrition in Adult Critically Ill Patients
Acronym: EPaNIC
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Greet Van den Berghe, MD PhD, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPaNIC 2007 1-2-2; ISRCTN 76223876; EudraCT 2007-000169-40; S 50404
Record Dates: First submitted 2007-07-31; First posted 2007-08-07 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness; Starvation
Keywords: early parenteral nutrition; critical illness; respiratory failure; kidney failure; hepatic failure; muscle strength; rehabilitation; overfeeding; Reduced Oral Intake
MeSH Terms: conditions — Critical Illness; Starvation; Hyperphagia; Respiratory Insufficiency; Renal Insufficiency; Liver Failure

STUDY DESIGN:
Who Masked: Investigator
Masking Description: All outcome adjudicators were unaware of study-group assignments
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EN only (Experimental): Withholding PN during the first week of ICU stay
  Interventions: Other: Withholding PN during the first week of ICU stay
- EN plus early PN (Active Comparator): Oliclinomel N71000 OR N71000E // Clinimix N17G35 OR N17G35E Parenteral nutrition targeted at covering calculated needs together with the enteral nutrition intake that is achieved
  Interventions: Drug: Oliclinomel N71000 OR N71000E // Clinimix N17G35 OR N17G35E

INTERVENTIONS:
Other: Withholding PN during the first week of ICU stay — Patients in this arm will receive exclusively enteral nutrition. If enteral nutrition is insufficient after the seventh day of ICU stay, parenteral nutrition will be started.
  Arms: EN only
Drug: Oliclinomel N71000 OR N71000E // Clinimix N17G35 OR N17G35E — PN will be started the morning of the third ICU hospitalisation day. The amount of PN to be given will be calculated to cover the caloric needs of the patient, based on the enteral energy intake the previous 24 hours.
  Other Names: Parenteral nutrition ATC code B05BA10
  Arms: EN plus early PN

SUMMARY:
In critically ill patients, a strategy aimed at an early delivery of full caloric support, with a combination of Enteral Nutrition (EN) and Parenteral Nutrition (PN) (in conditions preventing hyperglycemia and overfeeding), results in shorter ICU and hospital stay and less morbidity as compared to a strategy using only EN.

DETAILED DESCRIPTION:
Written informed consent will be obtained from the patient or the closest family member or legal guardian. The family member or the patient can withdraw from the trial, at any time, without impact on his treatment or penalty. The investigators confirm that this study concerns a condition that directly threatens patient health and that the adult patient not able to give consent suffers from the condition. The experiment is essential to confirm the results from earlier research in patients who could consent or from other research methods.

On admission patients will be randomly assigned to receive EN combined with early PN or only EN. At ICU admission, consecutive patients will be randomly assigned to one of these two treatment groups using blinded envelopes, stratified according to primary diagnostic category on admission. Upon addition of the new study site, the numbered en sealed envelopes for randomization stratified according to primary diagnostic category on admission were replaced by an identical digital system allowing central randomization.

As initial nutritional support, patients randomised to the 'EN combined with early PN' group will receive glucose 20% at 40 ml/hr. EN will be initiated in the evening of the second ICU hospitalisation day, PN will be started the morning of the third ICU hospitalisation day. The amount of PN to be given on any particular day will be the difference between calculated caloric needs and the calories delivered by EN the previous 24 hours. When EN covers 80% of calculated caloric needs PN will be stopped. When the patient is able to eat, the parenteral regimen will be reduced and eventually stopped. Whenever oral (+ enteral) intake is below 50% of calculated caloric needs, the PN will be (re)-started.

As initial nutritional support, patients randomised to the 'EN only' group will receive glucose 5% at 40 ml/hr. EN will be initiated on the evening of the second ICU day. From the morning of the third ICU hospitalisation day on, the amount of glucose 5% to be given will be the same as the volume of PN the patient theoretically would require to receive 100% of presumed caloric needs based on the amount of EN delivered the previous 24 hours. When the patient is able to eat, the parenteral regimen (glucose 5%) will be reduced to 50% and eventually stopped. Whenever oral (+ enteral) intake is below 50% of calculated caloric needs, the PN (glucose 5%) will be (re)-started. If these patients would need to stay for more than seven days on the ICU and enteral feeding of at least 80% of the calculated calories is not possible, they will be switched to EN and PN on day eight.

Common strategy for attempting early enteral nutrition in both study arms:

EN will be initiated on the evening of the second ICU day, unless patients are able to eat. The increase of enteral feeding volume and the adaptation of the regimen to pathological conditions will be according to protocol. Trace elements, minerals and vitamins will be administered daily intravenously (IV) to all patients from the day of admission onwards. IV substitution will be stopped in patients receiving at least 1500 ml of EN. All patients will be treated following the intensive insulin therapy schedule - targeting a blood glucose level of 80 - 110 mg/dl - from admission until discharge or oral feeding.

Patients will be weaned from the ventilator according to a standard protocol. End-of-care decisions in patients for whom further intensive care is considered to be futile will be taken in consensus by a group of two senior ICU physicians and the referring specialist, all blinded to study treatment allocation.

In a subgroup of patients, pathways of inflammation and metabolism and the endocrinological impact of the intervention will be studied in blood samples and in snap-frozen in vivo biopsies of muscle and adipose tissue. Blood and tissue samples from healthy volunteers will serve as references for these exploratory studies. In some patients, radiological evolution of regional muscle and adipose tissue volumes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to any of the five intensive care units
2. Older than 18 years
3. Nutritional risk screening score (NRS) higher or equal to three upon ICU admission

Exclusion Criteria:

1. Patients with a do not resuscitate (DNR) code or moribund at the time of ICU admission
2. Patients already enrolled in another trial
3. Patients transferred from another intensive care unit with an established nutritional therapy
4. Patients suffering from ketoacidotic or hyperosmolar coma on admission
5. Patients with a body mass index (BMI) below 17 kg/m^2
6. Short bowel syndrome
7. Patients known to be pregnant or nursing
8. Patients on mechanical ventilation at home
9. NRS score lower than three
10. Patient readmitted to ICU after randomization to the EPaNIC trial.
11. Patient not critically ill on admission. (No clinical indication for central intravenous catheter or patient ready for oral nutrition on admission.)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4640 (Actual)
Dates: Start 2007-08; Primary Completion 2011-02 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Length of stay in ICU and length of stay in the hospital. | 2 years

SECONDARY OUTCOMES:
Death (hospital and ICU mortality and 90 days mortality) | 10 years
Days to weaning from mechanical ventilation | 2 years
The need for renal replacement therapies | 2 years
The presence or absence of new kidney injury during intensive care | 2 years
Days of vasopressor or inotropic support | 2 years
The presence or absence of signs of ICU liver disease: hyperbilirubinemia (defined as bilirubin level > 3 mg/dl), presence of liversteatosis, sludge… | 2 years
The need for tracheotomy | 2 years
The presence or absence of hyper-inflammation within five days after ICU admission | 2 years
Blood lipid profiles and albumin on days one, five, ten, and fifteen after admission | 2 years
The presence or absence of bacteraemia, ventilator-associated pneumonia and of wound infections | 2 years
Episodes of hypoglycaemic events (defined as glycemia less than 40 mg/dl) | 2 years
Amount and type of calories delivered | 2 years
Muscle strength: among others: MRCss, Maximum Inspiratory Pressure in patients staying more than 7 days in ICU and a subset staying < 7 days, as well as in individuals who have never stayed in ICU. Presence of electrophysiological signs of CIP/CIM. | 10 years
Rehabilitation/functionality: among others: six minute walking distance and activities of daily life at hospital discharge and at follow-up moments. SF 36 questionnaire at several follow-up moments and in individuals who have never stayed in ICU. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Greet Van den Berghe, MD Ph D, Study Director — Director of the Department of Intensive Care Medicine Catholic Univeresity Leuven; Michaël P Casaer, MD, Principal Investigator — Department of Intensive Care Medicine Catholic University Leuven; Alexander P Wilmer, MD Ph D, Principal Investigator — Department of Medicine Catholic University Leuven; Jasperina Dubois, MD, Principal Investigator — Surgical Intensive Care Unit Regional Hospital Jessa
Locations (3):
- Belgium (3):
  - Surgical Intensive Care Unit Regional Hospital Jessa, Hasselt
  - Medical Intensive Care Unit, Leuven
  - Surgical Intensive Care Unit, Catholic University Leuven University Hospitals, Leuven

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Derived] Uzun Ayar C, Guiza F, Derese I, Pauwels L, Vander Perre S, Pintelon I, Casaer M, Van Aerde N, Hermans G, Derde S, Kreiss L, Van den Berghe G, Vanhorebeek I. Altered muscle transcriptome as molecular basis of long-term muscle weakness in survivors from critical illness. Intensive Care Med. 2025 Jun;51(6):1062-1077. doi: 10.1007/s00134-025-07949-3. Epub 2025 Jun 10. PMID 40493222
- [Derived] Casaer MP, Stragier H, Hermans G, Hendrickx A, Wouters PJ, Dubois J, Guiza F, Van den Berghe G, Gunst J. Impact of withholding early parenteral nutrition on 2-year mortality and functional outcome in critically ill adults. Intensive Care Med. 2024 Oct;50(10):1593-1602. doi: 10.1007/s00134-024-07546-w. Epub 2024 Jul 17. PMID 39017697
- [Derived] Van Dyck L, Guiza F, Derese I, Pauwels L, Casaer MP, Hermans G, Wouters PJ, Van den Berghe G, Vanhorebeek I. DNA methylation alterations in muscle of critically ill patients. J Cachexia Sarcopenia Muscle. 2022 Jun;13(3):1731-1740. doi: 10.1002/jcsm.12970. Epub 2022 Mar 11. PMID 35274472
- [Derived] Vanhorebeek I, Derese I, Gunst J, Wouters PJ, Hermans G, Van den Berghe G. Persisting neuroendocrine abnormalities and their association with physical impairment 5 years after critical illness. Crit Care. 2021 Dec 16;25(1):430. doi: 10.1186/s13054-021-03858-1. PMID 34915907
- [Derived] Ingels C, Langouche L, Dubois J, Derese I, Vander Perre S, Wouters PJ, Gunst J, Casaer M, Guiza F, Vanhorebeek I, Van den Berghe G. C-reactive protein rise in response to macronutrient deficit early in critical illness: sign of inflammation or mediator of infection prevention and recovery. Intensive Care Med. 2022 Jan;48(1):25-35. doi: 10.1007/s00134-021-06565-1. Epub 2021 Nov 24. PMID 34816288
- [Derived] Van Aerde N, Meersseman P, Debaveye Y, Wilmer A, Gunst J, Casaer MP, Wauters J, Wouters PJ, Gosselink R, Van den Berghe G, Hermans G. Five-year outcome of respiratory muscle weakness at intensive care unit discharge: secondary analysis of a prospective cohort study. Thorax. 2021 Jun;76(6):561-567. doi: 10.1136/thoraxjnl-2020-216720. Epub 2021 Mar 12. PMID 33712505
- [Derived] Van Dyck L, Gunst J, Casaer MP, Peeters B, Derese I, Wouters PJ, de Zegher F, Vanhorebeek I, Van den Berghe G. The clinical potential of GDF15 as a "ready-to-feed indicator" for critically ill adults. Crit Care. 2020 Sep 14;24(1):557. doi: 10.1186/s13054-020-03254-1. PMID 32928255
- [Derived] Van Aerde N, Meersseman P, Debaveye Y, Wilmer A, Gunst J, Casaer MP, Bruyninckx F, Wouters PJ, Gosselink R, Van den Berghe G, Hermans G. Five-year impact of ICU-acquired neuromuscular complications: a prospective, observational study. Intensive Care Med. 2020 Jun;46(6):1184-1193. doi: 10.1007/s00134-020-05927-5. Epub 2020 Jan 22. PMID 31970446
- [Derived] Hermans G, Van Aerde N, Meersseman P, Van Mechelen H, Debaveye Y, Wilmer A, Gunst J, Casaer MP, Dubois J, Wouters P, Gosselink R, Van den Berghe G. Five-year mortality and morbidity impact of prolonged versus brief ICU stay: a propensity score matched cohort study. Thorax. 2019 Nov;74(11):1037-1045. doi: 10.1136/thoraxjnl-2018-213020. Epub 2019 Sep 3. PMID 31481633
- [Derived] Van Dyck L, Derese I, Vander Perre S, Wouters PJ, Casaer MP, Hermans G, Van den Berghe G, Vanhorebeek I. The GH Axis in Relation to Accepting an Early Macronutrient Deficit and Outcome of Critically Ill Patients. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5507-5518. doi: 10.1210/jc.2019-00842. PMID 31361307
- [Derived] Thiessen SE, Derde S, Derese I, Dufour T, Vega CA, Langouche L, Goossens C, Peersman N, Vermeersch P, Vander Perre S, Holst JJ, Wouters PJ, Vanhorebeek I, Van den Berghe G. Role of Glucagon in Catabolism and Muscle Wasting of Critical Illness and Modulation by Nutrition. Am J Respir Crit Care Med. 2017 Nov 1;196(9):1131-1143. doi: 10.1164/rccm.201702-0354OC. PMID 28475354
- [Derived] Flechet M, Guiza F, Schetz M, Wouters P, Vanhorebeek I, Derese I, Gunst J, Spriet I, Casaer M, Van den Berghe G, Meyfroidt G. AKIpredictor, an online prognostic calculator for acute kidney injury in adult critically ill patients: development, validation and comparison to serum neutrophil gelatinase-associated lipocalin. Intensive Care Med. 2017 Jun;43(6):764-773. doi: 10.1007/s00134-017-4678-3. Epub 2017 Jan 27. PMID 28130688
- [Derived] Hermans G, Van Mechelen H, Bruyninckx F, Vanhullebusch T, Clerckx B, Meersseman P, Debaveye Y, Casaer MP, Wilmer A, Wouters PJ, Vanhorebeek I, Gosselink R, Van den Berghe G. Predictive value for weakness and 1-year mortality of screening electrophysiology tests in the ICU. Intensive Care Med. 2015 Dec;41(12):2138-48. doi: 10.1007/s00134-015-3979-7. Epub 2015 Aug 13. PMID 26266842
- [Derived] Hermans G, Van Mechelen H, Clerckx B, Vanhullebusch T, Mesotten D, Wilmer A, Casaer MP, Meersseman P, Debaveye Y, Van Cromphaut S, Wouters PJ, Gosselink R, Van den Berghe G. Acute outcomes and 1-year mortality of intensive care unit-acquired weakness. A cohort study and propensity-matched analysis. Am J Respir Crit Care Med. 2014 Aug 15;190(4):410-20. doi: 10.1164/rccm.201312-2257OC. PMID 24825371
- [Derived] Hermans G, Casaer MP, Clerckx B, Guiza F, Vanhullebusch T, Derde S, Meersseman P, Derese I, Mesotten D, Wouters PJ, Van Cromphaut S, Debaveye Y, Gosselink R, Gunst J, Wilmer A, Van den Berghe G, Vanhorebeek I. Effect of tolerating macronutrient deficit on the development of intensive-care unit acquired weakness: a subanalysis of the EPaNIC trial. Lancet Respir Med. 2013 Oct;1(8):621-629. doi: 10.1016/S2213-2600(13)70183-8. Epub 2013 Sep 10. PMID 24461665
- [Derived] Boonen E, Vervenne H, Meersseman P, Andrew R, Mortier L, Declercq PE, Vanwijngaerden YM, Spriet I, Wouters PJ, Vander Perre S, Langouche L, Vanhorebeek I, Walker BR, Van den Berghe G. Reduced cortisol metabolism during critical illness. N Engl J Med. 2013 Apr 18;368(16):1477-88. doi: 10.1056/NEJMoa1214969. Epub 2013 Mar 19. PMID 23506003
- [Derived] Langouche L, Vander Perre S, Marques M, Boelen A, Wouters PJ, Casaer MP, Van den Berghe G. Impact of early nutrient restriction during critical illness on the nonthyroidal illness syndrome and its relation with outcome: a randomized, controlled clinical study. J Clin Endocrinol Metab. 2013 Mar;98(3):1006-13. doi: 10.1210/jc.2012-2809. Epub 2013 Jan 24. PMID 23348400
- [Derived] Casaer MP, Wilmer A, Hermans G, Wouters PJ, Mesotten D, Van den Berghe G. Role of disease and macronutrient dose in the randomized controlled EPaNIC trial: a post hoc analysis. Am J Respir Crit Care Med. 2013 Feb 1;187(3):247-55. doi: 10.1164/rccm.201206-0999OC. Epub 2012 Nov 29. PMID 23204255
- [Derived] Vanderheyden S, Casaer MP, Kesteloot K, Simoens S, De Rijdt T, Peers G, Wouters PJ, Coenegrachts J, Grieten T, Polders K, Maes A, Wilmer A, Dubois J, Van den Berghe G, Mesotten D. Early versus late parenteral nutrition in ICU patients: cost analysis of the EPaNIC trial. Crit Care. 2012 May 25;16(3):R96. doi: 10.1186/cc11361. PMID 22632574
- [Derived] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Derived] Casaer MP, Hermans G, Wilmer A, Van den Berghe G. Impact of early parenteral nutrition completing enteral nutrition in adult critically ill patients (EPaNIC trial): a study protocol and statistical analysis plan for a randomized controlled trial. Trials. 2011 Jan 24;12:21. doi: 10.1186/1745-6215-12-21. PMID 21261975
- See also: Katholieke Universiteit Leuven Homepage — https://gbiomed.kuleuven.be/english/research/50000618/50000663/
- See also: Casaer et al.: Impact of early parenteral nutrition completing enteral nutrition in adult critically ill patients (EPaNIC trial): a study protocol and statistical analysis plan for a randomized controlled trial. Trials 2011 12:21. — http://www.trialsjournal.com/content/12/1/21/abstract
- See also: Casaer MP et al.: Early versus late parenteral nutrition in critically ill adults — http://www.nejm.org/doi/full/10.1056/NEJMoa1102662